CLINICAL TRIAL: NCT02636400
Title: Is Postoperative IUI Better Than Expectant Management in Infertile Endometriosis Patients With Good Prognosis Based on EFI Score?
Brief Title: Immediate Intra Uterine Isemination (IUI) Versus Expectant Management in Postoperative Endometriosis Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted prematurely
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S55983
Record Dates: First submitted 2015-03-23; First posted 2015-12-21 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Endometriosis; Infertility
Keywords: Infertility; endometriosis
MeSH Terms: conditions — Endometriosis; Infertility | interventions — Gonadotropins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- expectant (No Intervention): 7 menstrual cycles of expectant management
- postop IUI (Experimental): 4 IUI cycles within 7 menstrual cycles
  Interventions: Other: controlled ovarian stimulation with gonadotropins + intrauterine insemination

INTERVENTIONS:
Other: controlled ovarian stimulation with gonadotropins + intrauterine insemination
  Other Names: postop IUI
  Arms: postop IUI

SUMMARY:
Is postoperative IUI better than expectant management in infertile endometriosis patients with good prognosis based on their EFI score? (A single centre randomised controlled trial).

ELIGIBILITY:
Inclusion Criteria:

* recent (<6months) complete laparoscopic endometriosis resection
* endometriosis fertility index (EFI) at least 7/10
* Regular menstrual cycles (min 24days - max 38days) with proven ovulation
* At least one functional tube at surgery, normal uterus
* Sperm sample of partner: normal or mild male factor

Exclusion Criteria:

* frozen (donor or partner) sperm
* clinical and/or imaging evidence of endometriosis recurrence/persistence at randomization
* FSH > 20 IU/L

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
cumulative clinical pregnancy rate | participants will be followed for the duration of 7 menstrual cycles and in case of pregnancy, they will be followed until the pregnancy outcome is known, implying an average time frame of 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D'Hooghe, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium